CLINICAL TRIAL: NCT05939232
Title: Registry of X-linked Adrenoleukodystrophy
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Other Study IDs: KY2023-011-02
Record Dates: First submitted 2023-05-16; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: X-linked Adrenoleukodystrophy
Keywords: X-linked Adrenoleukodystrophy; Genetic data; Phenotype; Imaging feature; Mechanism
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood, urine, and feces were retained at baseline, 1 year, 2 year, 3 year, 4 year and 5 year during follow-up. Details of biospecimen sampling as the following:
  numbers of sampling: 200 subjects; serum: 21600 tubes, 0.5mL/tube; plasma: 7200 tubes, 0.5mL/tube; urine: 24000 tubes, 1mL/tube; feces: 7200 tubes, 12g/tube; other biospecimen (white blood cell): 6000 tubes, 0.5mL/tube.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- X-ALD: X-linked adrenoleukodystrophy (X-ALD) patients.
- Carrier-control (CC): Carriers of mutation in gene encoding ATP-binding cassette subfamily D member 1 (ABCD1), who have no X-linked adrenoleukodystrophy and are matched with the X-ALD group according to age, sex and education.

SUMMARY:
This study is a observational study conducted through recruiting X-linked adrenoleukodystrophy (X-ALD) patients, to build a comprehensive evaluation and long-term follow-up platform for X-ALD patients, and to provide a theoretical basis for the treatment and management of X-ALD patients.

DETAILED DESCRIPTION:
In this study, X-ALD patients will be selected as study participants. Through a longitudinal collection of genetic, imaging and clinical symptoms data of the patients and carriers. The purpose of this study is to build a comprehensive evaluation and long-term follow-up platform for X-ALD patients. Through the long-term follow-up of imaging and clinical symptoms progress and outcome of X-ALD patients, combined with genetic data, we will improve the relationships between genes and phenotypes, and explore the deep insight in the pathophysiological mechanism of X-ALD, to provide a theoretical basis for the treatment and management of X-ALD patients.

ELIGIBILITY:
Inclusion Criteria:

X-ALD group：

* Meet the diagnostic criteria of X-ALD and supported by the results of genetic and very long chain fatty acid (VLCFA) test;
* Age: 6 - 70 years old;
* Able to communicate normally, and complete the test of scale as instructed (confirmed by the field test of scale);
* Sign the informed consent.

Carrier-control group:

Healthy people who have no significant difference in age, sex and education comparing with the X-ALD group, volunteer to participate in this study, could complete the test of scale as instructed, and meet the following criteria:

* Eligible for asymptomatic carriers in genetic tests (preference of patient's mother and close relatives);
* Age: 6 - 70 years old, able to complete the test of scale as instructed (confirmed by the field test of scale);
* No history of psychiatric diseases.

Exclusion Criteria:

* Other hereditary diseases;
* Other severe central nervous diseases;
* History of surgery of brain or eye;
* Psychiatric and psychological diseases, such as anxiety and depression;
* Metal foreign body or prosthesis in the human body (such as pacemaker and insulin pump), claustrophobia, and other MRI contraindications;
* History of surgery associated with gastrointestinal tract;
* No informed consent;
* Unable to tolerate MRI or eye related tests.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: X-linked adrenoleukodystrophy patients, and age,sex and education matched healthy carriers will be recruited from the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Epidemiological characteristics in Chinese X-ALD patients | 5 years
  Constructing a Chinese X-ALD epidemiological information database by collecting epidemiological information from X-ALD patients.
Clinical characteristics in Chinese X-ALD patients | 5 years
  Constructing a Chinese X-ALD clinical sympotoms information database by collecting clinical symptoms information from X-ALD patients.
Imaging characteristics in Chinese X-ALD patients | 5 years
  Constructing a Chinese X-ALD patient's head MRI information database by collecting head MRI information from X-ALD patients.
The disease development in Chinese X-ALD patients | 5 years
  Record the progress of patients' clinical symptoms from baseline through 5-year follow-up.
New pathogenic loci of Chinese X-ALD patients in whole genome sequencing/whole exon sequencing | 5 years
  To find and identify new pathogenic loci of X-ALD in whole genome sequencing/whole exon sequencing through comparing the differences of whole genome sequencing/whole exon sequencing between X-ALD patients and carrier-control individuals.

SECONDARY OUTCOMES:
Etiology of Chinese X-ALD patients | 5 years
  Etiological factors,including genetic and environmental etiological factors, will be explored by genomic analysis, lasso regression, multiple logistic regression, and cox proportional hazards regression.
The change of imagin features in Chinese X-ALD patients | day 1, year 1, year 2, year 3, year 4, year 5
  Record the change of the patient's head MRI from baseline through follow-up every year.
The associations between genetic factors and clinical characteristics of Chinese X-ALD patients | 5 years
  β coefficient and 95%CI values in linear regression, OR and 95%CI values in logistic regression analysis, and HR and 95%CI values in cox proportional hazards regression analysis for the associations between genetic factors and clinical characteristics of X-ALD.
The associations between genetic factors and outcomes of Chinese X-ALD patients | 5 years
  β coefficient and 95%CI values in linear regression, OR and 95%CI values in logistic regression analysis, and HR and 95%CI values in cox proportional hazards regression analysis for the associations between genetic factors and outcomes of X-ALD.
The associations between genetic factors and imaging characteristics of Chinese X-ALD patients | 5 years
  β coefficient and 95%CI values in linear regression, OR and 95%CI values in logistic regression analysis, and HR and 95%CI values in cox proportional hazards regression analysis for the associations between genetic factors and imaging characteristics of X-ALD.
The associations between genetic factors and the long-term changes of imaging characteristics of Chinese X-ALD patients | 5 years
  β coefficient and 95%CI values in linear regression, OR and 95%CI values in logistic regression analysis, and HR and 95%CI values in cox proportional hazards regression analysis for the associations between genetic factors and the long-term changes of imaging characteristics of X-ALD.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, MD,PhD, Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tiantan Hospital, Beijing, China